CLINICAL TRIAL: NCT06155513
Title: Impact of a Daily Application of Omega-3 Monoglycerides Based Serum and Cream on Self-assessment of Eczema Severity as Well as on the Ratio of 4 Bacteria of the Skin Microbiota (Staphylococcus Aureus, Staphylococcus Epidermis, Cutibacterium Acnes and Streptococcus Pyogenes): Exploratory Study (COS-PBP-02)
Brief Title: Omega-3 Monoglyceride Based Topic Products as Skin Prebiotics for Eczema
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SCF Pharma (Industry)
Collaborators: Institut de recherche clinique du littoral (IRCL) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: COS-PBP-02
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Eczema
Keywords: Skin hydration; Skin inflammation
MeSH Terms: conditions — Eczema; Dermatitis | interventions — Light

STUDY DESIGN:
Intervention Model Description: This exploratory study includes two groups of eight (8) subjects. Subjects of group A will receive treatment A (serum A and cream A). Subjects of group B will receive treatment B (serum B and cream B). A skin area with eczema lesions will be identified during the screening visit. Subjects will be asked to apply the serum, then the cream to the targeted area at least once a day for a period of forty-two (42) days. The pre-treatment baseline state will serve as a control for the effects observed following treatment on the targeted area.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Serum and Cream of formulation A (light) (Experimental): Daily application of glyceryl Eicosapentaenoate serum and glyceryl Eicosapentaenoate cream of formulation A on the targeted skin area. The skin area must be clean and dry. Subjects must proceed with at least one application of products each day for 42 consecutive days. Subjects may proceed with additional daily product applications if needed.
  Interventions: Combination Product: Omega-3 monoglyceride based topical Serum and cream of formulation A (light)
- Group B: Serum and Cream of formulation B (rich) (Experimental): Daily application of glyceryl Eicosapentaenoate serum and glyceryl Eicosapentaenoate cream of formulation B on the targeted skin area. The skin area must be clean and dry. Subjects must proceed with at least one application of products each day for 42 consecutive days. Subjects may proceed with additional daily product applications if needed.
  Interventions: Combination Product: Omega-3 monoglyceride based topical Serum and cream of formulation B (rich)

INTERVENTIONS:
Combination Product: Omega-3 monoglyceride based topical Serum and cream of formulation A (light) — Omega-3 monoglyceride based serum and cream of lighter formulation
  Other Names: Serum and cream of formulation A (light)
  Arms: Group A: Serum and Cream of formulation A (light)
Combination Product: Omega-3 monoglyceride based topical Serum and cream of formulation B (rich) — Omega-3 monoglyceride based serum and cream with a richer formulation
  Other Names: Serum and cream of formulation B (rich)
  Arms: Group B: Serum and Cream of formulation B (rich)

SUMMARY:
This exploratory study aims to verify the impact on the severity of eczema as well as the prebiotic potential of a daily application of Omega-3 serum and cream on a skin with eczema. This study will also collect data on possible adverse effects of the products. Sixteen participants will be enrolled in this study and will be divided in two groups of 8 subjects that will receive two different treatments for forty-two days. The baseline condition will serve as a control for the effects observed after treatment on the targeted eczema area.

DETAILED DESCRIPTION:
Omega-3 fatty acids and more particularly EPA are recognized as fatty acids promoting the resolution of inflammation unlike omega-6 fatty acids, which are pro-inflammatory. The skin, which is the largest organ of the human body, receives a greater proportion of omega-6 fatty acids because skin care products are mostly made of omega-6-rich vegetable oil. This imbalance could be one of the causes of inflammatory skin diseases such as eczema. Conventional omega-3 need to pass through the digestive tract to be activated in the form of monoglycerides. Hence, it is not relevant to use them for a topical formulation. However, the recent development of pre-activated omega-3 monoglycerides finally opens the possibility of introducing active omega-3 fatty acids into moisturizing products.

Subjects of group A will receive treatment A coinsisting of serum A and cream A. Subjects of group B will receive treatment B coinsisting of serum B and cream B. A skin area with eczema lesions will be identified during the screening visit. Subjects will be asked to apply the provided serum and cream to the clean targeted area at least once a day, every day, for a period of forty-two (42) days. The pre-treatment baseline state will serve as a control for the effects observed following treatment on the targeted area.

The targeted eczema area will be used to measure the main parameters of the study:

1. Quantify by qPCR the four main bacteria of the skin microbiota (Staphylococcus aureus, Staphylococcus epidermis, Cutibacterium acnes and Streptococcus pyogenes). Specimens will be collected before the start of treatment (visit 1) as well as after three weeks (visit 2) and six weeks of treatment (visit 3).
2. Compare the evolution of eczema lesions pre and post treatment by administering a self-assessment questionnaire for eczema severity (POEM). The POEM questionnaire will be administered before the start of treatment (visit 1) as well as after three weeks (visit 2) and six weeks of treatment (visit 3).

This study will also aim to collect data on the possible undesired effects of the products.

ELIGIBILITY:
Inclusion Criteria:

1. Participant aged of at least 18 years old.
2. Participant diagnosed with eczema who did not use corticosteroids in the 14 days prior to study day 1;
3. Available for the entire duration of the study and willing to participate based on the information provided in the ICF duly read and signed by the latter.
4. Participant without intellectual problems likely to limit the validity of consent to participate in the study and compliance with protocol requirements, having the ability to cooperate adequately, understand and observe the instructions of research staff.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Impact of treatment on participant's self-assessment of eczema severity | 6 weeks
  Participants will be asked to complete a self-assessment eczema questionnaire (Patient Oriented Eczema Measure - POEM) before the start of treatment and after three (3) and six (6) weeks of treatment. The POEM score will determine eczema severity. The score ranges from 0 to 28: 0 being a normal skin, 3 to 7 is a mild eczema, 8 to 16 is moderate, 17 to 24 in severe and 25 to 28 is very severe eczema.
Quantification by qPCR of the four main bacteria of the skin microbiota at the targeted eczema zone. | 6 weeks
  A specimen of the skin microbiota at the targeted eczema area will be taken by swab before the start of treatment as well as after three (3) and six (6) weeks of treatment. The specimens will be analyzed by qPCR targeting the genome of four bacteria: Staphylococcus aureus, Staphylococcus epidermis, Cutibacterium acnes and Streptococcus pyogenes.

SECONDARY OUTCOMES:
Assessment of potential adverse effects of treatment | 6 weeks
  At each study visit and follow-ups, subjects will be questioned for any change in the health of the treated skin area. They will also be asked to report any adverse effects observed on the treated area for each period inbetween visits.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel P Fortin, Ph.D, Principal Investigator — SCF Pharma
Locations (1):
- SCF Pharma, Rimouski, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
The results of this research are the private property of SCF Pharma. If you are interested in the results of this study, you can contact Dr Samuel Fortin for a summary starting in summer 2025.

REFERENCES:
- [Background] Simopoulos AP. The importance of the ratio of omega-6/omega-3 essential fatty acids. Biomed Pharmacother. 2002 Oct;56(8):365-79. doi: 10.1016/s0753-3322(02)00253-6. PMID 12442909
- [Background] Costantini L, Molinari R, Farinon B, Merendino N. Impact of Omega-3 Fatty Acids on the Gut Microbiota. Int J Mol Sci. 2017 Dec 7;18(12):2645. doi: 10.3390/ijms18122645. PMID 29215589
- [Background] Koh LF, Ong RY, Common JE. Skin microbiome of atopic dermatitis. Allergol Int. 2022 Jan;71(1):31-39. doi: 10.1016/j.alit.2021.11.001. Epub 2021 Nov 24. PMID 34838450
- [Background] Purnamawati S, Indrastuti N, Danarti R, Saefudin T. The Role of Moisturizers in Addressing Various Kinds of Dermatitis: A Review. Clin Med Res. 2017 Dec;15(3-4):75-87. doi: 10.3121/cmr.2017.1363. Epub 2017 Dec 11. PMID 29229630